CLINICAL TRIAL: NCT06014034
Title: Randomized Controlled Study of Programmed Weaning From Noninvasive Mechanical Ventilation for Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Randomized Controlled Study of Programmed Weaning From NIV for AECOPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y75505-04
Record Dates: First submitted 2023-08-09; First posted 2023-08-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Acute Exacerbation of COPD
Keywords: noninvasive mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Programmed Weaning From Noninvasive Mechanical Ventilation
  Interventions: Other: Programmed Weaning From Noninvasive Mechanical Ventilation
- Control group (No Intervention): this is the traditional withdrawal unit (the attending physician will decide the NIV regimen according to the condition).

INTERVENTIONS:
Other: Programmed Weaning From Noninvasive Mechanical Ventilation — Programmed withdrawal unit: daily morning review arterial blood gas analysis (since the 2nd, daily morning stop non-invasive ventilation 1 hours, 2 hours, 3 hours, 4 hours after check arterial blood gas analysis), blood gas results suggest respiratory acidosis compensatory period (pH value greater than 7.35) can reduce daily noninvasive ventilation time, namely the noninvasive ventilation use time for 24 hours, 20 hours, the third day 16 hours, the fourth 12 hours, fifth day 8 hours. If ABG indicates still acid decompensation, continue the non-invasive ventilation regimen of the previous day. If noninvasive ventilation failed, invasive mechanical ventilation was performed.
  Arms: Study group

SUMMARY:
Purpose of research:to explore a reasonable programmed withdrawal process of noninvasive ventilation and thereby reduce the duration of noninvasive mechanical ventilation in patients with acute exacerbations of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized controlled study. The study subjects were patients with acute exacerbation of chronic obstructive pulmonary disease admitted to the intensive care unit, who were randomized into the study group, that is, the programmed withdrawal unit, and the control group was the traditional withdrawal unit (the attending physician decided the NIV regimen according to the condition). The primary study endpoints of the trial were complete evacuation of noninvasive ventilation (i. e. from the start of the patient to noninvasive ventilation) or return of time to normal ventilation for patients with a home non-invasive ventilator prior to acute exacerbation. Secondary study endpoints include length of stay, stay and failure of non-invasive ventilation (failure of non-invasive ventilation was defined as the patient requiring endotracheal intubation to invasive ventilation or death).

ELIGIBILITY:
Inclusion Criteria:

* It is defined that in patients with acute exacerbation of chronic obstructive pulmonary disease, the arterial blood gas analysis was decompensation of respiratory acidosis, and the pH value was 7.20-7.35
* Non-invasive mechanical ventilation was performed and it was well tolerated

Exclusion Criteria:

* younger than 40 years old
* pregnancy
* Human immunodeficiency virus (HIV) antibody was positive
* Hemodynamic instability
* Mechanical ventilation for endotracheal intubation and cardiopulmonary resuscitation were disagreed

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete evacuation time of non-invasive ventilation | At the end of non-invasive ventilation，through study completion, an average of 11 days
  from the start of the patient to the absence of noninvasive ventilation or return to the level of normal ventilation time for patients with non-invasive ventilation on a home non-invasive ventilator before acute exacerbation

SECONDARY OUTCOMES:
Time in the ICU | At the end of therapy in ICU，through study completion, an average of 14 days
  from the start of the patient stay in ICU to the day leave from ICU
length of stay | At the end of therapy in hospital, through study completion, an average of 20 days
  from the start of the patient stay in hospital to leave from hospital
Failure rate of non-invasive ventilation | At the end of therapy in hospital, an average of 20 days
  failure of non-invasive ventilation is defined as a patient requiring endotracheal intubation to invasive ventilation or death

CONTACTS AND LOCATIONS:
Overall Officials: Qingtao Zhou, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospita, Beijing, Beijing Municipality, China